CLINICAL TRIAL: NCT04766697
Title: An Integrated Substance Use, Violence, and HIV/AIDS Syndemic Risk-reduction Intervention for African American Couples
Brief Title: SAVA Syndemic Risk Reduction for African American Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5R03DA044866-02 (NIH)
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: SAVA
Keywords: HIV, couples, IPV, substance abuse, African American
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receive Intervention (Experimental): All 20 couples will receive the 8-session adapted intervention.
  Interventions: Behavioral: Risk-Reduction Sessions

INTERVENTIONS:
Behavioral: Risk-Reduction Sessions — The 8-session intervention protocol emphasizes cognitive-behavioral interventions for anger management, conflict resolution, reducing sexual risk behavior, substance use, and enhancement of couple functioning.

SUMMARY:
Synergistic interactions among substance abuse, violence, and HIV/AIDS, dubbed the SAVA syndemic, are highly linked to HIV acquisition among African Americans. Given limited literature and development of interventions for HIV-negative but high-risk heterosexual AA couples, there is a need for SAVA risk-reduction development tailored to this population. Phase 1 consisted of qualitative interviews with 16 couples who met study criteria to gather input and information to adapt an 8-session couple-based SAVA syndemic informed risk reduction intervention for HIV-negative, AA heterosexual couples who reported intimate partner violence (IPV) and substance abuse. Phase 2 is the focus of this trial and will consist of delivery of the intervention to 20 couples who meet study inclusion criteria to test the adapted intervention. Given the disproportionate impact of HIV on AAs, this study addresses a key gap in literature by testing the first SAVA informed risk-reduction intervention for high-risk, HIV-negative, heterosexual AA couples.

DETAILED DESCRIPTION:
Synergistic interactions between substance use, violence, and HIV/AIDS (SAVA syndemic) are closely linked with HIV acquisition among African Americans (AAs). However, no interventions have been developed to address SAVA syndemic risk-reduction for HIV-negative but high-risk heterosexual AA couples. This application builds on a qualitative study that was conducted during phase 1 of a NIDA-funded project. In phase 1, the investigators finalized and tested our recruitment protocol and conducted qualitative interviews with 16 couples who met study criteria. This application focused on phase 2 of the funded study. As part of this study the investigators will test an adapted 8-session couple-based SAVA syndemic informed risk-reduction intervention for HIV-negative, AA heterosexual couples who report intimate partner violence (IPV), and substance use. For this purpose, the investigators deliver the intervention to 20 couples who meet study inclusion criteria to test the adapted intervention. The intervention will be delivered online (via zoom) to individual couples. These couples will be recruited through social media (Facebook, Instagram, and Twitter) and advertising through local community-based organizations. The investigators will also inform the couples who participated in phase 1 qualitative interviews about the opportunity to participate in phase 2. Those who express an interest in participating in phase 2 will have to complete screening again to make sure they are eligible for the present study. This research will be done as part of a grant proposal funded by NIDA. Given the disproportionate impact of HIV on AAs, this study addresses a key gap in literature by testing the first SAVA informed risk-reduction intervention for high-risk, HIV-negative, heterosexual AA couples.

ELIGIBILITY:
Inclusion Criteria:

Both participants must:

* be between 18-49 years old
* self-identify as African American/Black
* identify each other as the main/steady heterosexual partner
* have been together for at least 2 months
* plan to be together for at least 3 months
* have had unprotected anal/ vaginal sex with their partner in the last 3 months.

At least one participant must have engaged in:

* IPV in the relationship in the last 6 months
* substance use in the last 6 months.

Exclusion Criteria:

* <18 or >49 years of age
* not being African American/ Black
* not having a steady partner of the opposite sex for at least 2 months
* not sexually active in the last 3 months
* currently pregnant or planning a pregnancy in the next 6 months
* not English language proficient
* showing evidence of significant cognitive impairment at screening; and (h) reporting severe physical or sexual violence by partner in the last 6 months (required medical attention) or being fearful of the partner.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Condom use | 2-months
  frequency of protected and unprotected vaginal and anal sex
Attitudes toward Sexual Partner Concurrency | 2-months
  10-item self-report measure of attitudes toward sexual partner concurrency
Intimate Partner Violence | 2-months
  38-items Conflict Tactics Scale measures victimization and perpetration of physical, psychological, and sexual violence
Drug use | 2-months
  10-item Drug Abuse Screening Test (DAST-10) will be used to assess changes in drug use

SECONDARY OUTCOMES:
Mental Health | 2-months
  PHQ-9 will be used to assess depressive symptoms
Relationship Satisfaction | 2-months
  Couple Satisfaction Index (CSI-16) will be used to assess relationship satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mittal, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland School of Public Health, Department of Family Sciences, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No